CLINICAL TRIAL: NCT01175616
Title: Creatine Augmentation in Female & Male Veterans With Selective Serotonin Reuptake Inhibitor-Resistant Major Depressive Disorder
Brief Title: Creatine Augmentation in Veterans With SSRI-Resistant Major Depression
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study withdrawn from ClinicalTrials.gov.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Douglas Kondo, MD, MD, University of Utah
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00041936
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Adults
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Creatine (Experimental): Open-Label Active Treatment with Creatine 5 grams daily for 8 weeks.
  Interventions: Drug: Creatine

INTERVENTIONS:
Drug: Creatine — Oral Creatine 5 grams daily.
  Other Names: Creapure

SUMMARY:
The purpose of this study is to determine whether creatine will be helpful as an adjunctive treatment for treatment-resistant major depressive disorder (MDD) in female and male Veterans. We hypothesize that Veterans receiving creatine will show decreased depressive symptoms as measured by the Montgomery-Asberg Depression Rating Scale (MADRS). We will also use 31-Phosphorus Magnetic Resonance Spectroscopy (31-P MRS) brain scans to compare levels of neurochemicals related to energy metabolism in the brain, before-and-after treatment with creatine, and between healthy controls and MDD participants.

DETAILED DESCRIPTION:
This is an open-label clinical trial of the investigational drug creatine for augmentation treatment of female and male Veterans, ages 18-55, with Major Depressive Disorder (MDD) who have failed to respond to antidepressant treatment with a selective serotonin reuptake inhibitor (SSRI) drug. Based on converging preclinical and animal model research, and our laboratory's prior clinical trials, we hypothesize that the nutritional supplement creatine may provide benefit as an adjunctive treatment to SSRI pharmacotherapy, for Veterans with treatment-resistant depression.

Twenty (n=20) Veterans between the ages of 18-55 years with MDD will be recruited for participation in an open-label trial of creatine augmentation. Veterans with depression will have unremitted MDD, despite having had an adequate trial of an SSRI antidepressant. Participants with MDD will be treated with oral creatine 5 gm daily for 8 weeks and will continue taking their SSRI antidepressant. Participants will undergo brain scanning at baseline, and the scans will be repeated following 8 of adjunctive creatine.

The neuroimaging technique utilized is Phosphorus-31 Magnetic Resonance Spectroscopy (31P-MRS). 31P-MRS is a non-invasive method with no exposure to ionizing radiation. At the magnetic field strength utilized (3 Tesla), magnetic resonance imaging is FDA-approved and is not associated with irreversible or serious adverse events. Furthermore, 31P-MRS is the only in vivo method for in vivo quantification of phosphorus energy metabolism, in living human brain.

In addition to Veterans with MDD, twenty (n=20) healthy control (HC) participants will be recruited. HCs will be Veterans between the ages of 18-55, who have no history of psychiatric or substance use disorder. No treatment will be administered to HC participants.

The HCs will undergo a single 31P-MRS scan, which will be used to measure the phosphorus-bearing neurometabolites that are involved in brain energy metabolism. The research team will use data from 31P-MRS scans to compare levels of high-energy phosphate metabolites in MDD participants vs. healthy controls.

In addition, comparison of pre- and post-treatment 31P-MRS metabolite levels will be conducted in the MDD participants, to test the hypothesis that creatine augmentation improves brain energy metabolism.

ELIGIBILITY:
Inclusion Criteria for Major Depressive Disorder Participants:

* Must be a U.S. military Veteran from 18-55 years of age.
* Must meet DSM criteria for Major Depressive Disorder (MDD).
* Current depressive episode duration of 4 weeks or longer.
* Montgomery-Asberg Depression Rating Scale (MADRS) score of 18 or greater.
* Adequate trial of an SSRI antidepressant, in terms of dosing and duration.
* No change in SSRI dose, for 4 weeks prior to the baseline brain scan.
* Partial or non-responder to current SSRI pharmacotherapy.

Exclusion Criteria for Major Depressive Disorder Participants:

* Primary psychotic or schizophrenia-spectrum disorder.
* Unstable co-morbid medical, neurologic, or psychiatric illness.
* Clinically significant substance use disorder.
* Significant risk of suicide, in the clinical judgment of the study physician.
* Inability to provide informed consent.
* Contraindication to brain scanning (e.g., pacemaker, ferromagnetic implant).
* Pre-existing renal disease, with proteinuria at baseline.
* History of hypersensitivity to creatine.
* Concurrent participation in another FDA-sanctioned clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) Score | screening; baseline; weeks 1, 2, 4, 5, 8, and 10
  The primary clinical outcome measure will be the change in MADRS; response will be defined as a 50% or greater decrease in MADRS score from baseline and a Clinical Global Impression Scale (CGI) improvement score of 1 or 2

SECONDARY OUTCOMES:
Changes in 3T 31Phosphorus Magnetic Resonance Spectroscopy metabolites | Baseline and 8 weeks
  The primary neuroimaging outcome measures will be changes in 3T 31P-MRS metabolites (PCr and β-NTP) globally and in the anterior cingulate cortex

CONTACTS AND LOCATIONS:
Overall Officials: Perry F Renshaw, MD, PhD, MBA, Study Director — University of Utah

IPD SHARING:
Plan to Share IPD: No
The study was closed prior to human subjects receiving investigational treatment.

REFERENCES:
- [Background] Lyoo IK, Yoon S, Kim TS, Hwang J, Kim JE, Won W, Bae S, Renshaw PF. A randomized, double-blind placebo-controlled trial of oral creatine monohydrate augmentation for enhanced response to a selective serotonin reuptake inhibitor in women with major depressive disorder. Am J Psychiatry. 2012 Sep;169(9):937-945. doi: 10.1176/appi.ajp.2012.12010009. PMID 22864465
- [Background] Kondo DG, Sung YH, Hellem TL, Fiedler KK, Shi X, Jeong EK, Renshaw PF. Open-label adjunctive creatine for female adolescents with SSRI-resistant major depressive disorder: a 31-phosphorus magnetic resonance spectroscopy study. J Affect Disord. 2011 Dec;135(1-3):354-61. doi: 10.1016/j.jad.2011.07.010. Epub 2011 Aug 9. PMID 21831448
- [Background] Allen PJ, D'Anci KE, Kanarek RB, Renshaw PF. Sex-specific antidepressant effects of dietary creatine with and without sub-acute fluoxetine in rats. Pharmacol Biochem Behav. 2012 Jun;101(4):588-601. doi: 10.1016/j.pbb.2012.03.005. Epub 2012 Mar 10. PMID 22429992
- [Background] Allen PJ. Creatine metabolism and psychiatric disorders: Does creatine supplementation have therapeutic value? Neurosci Biobehav Rev. 2012 May;36(5):1442-62. doi: 10.1016/j.neubiorev.2012.03.005. Epub 2012 Mar 24. PMID 22465051
- See also: Research Website - University of Utah Brain Instititue — http://www.utahbrain.org